CLINICAL TRIAL: NCT06743854
Title: Predisposing Factors for Liver Diseases in Patients With Chronic Hemolytic Anemia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Saadiea Abdo Bedir Eid, Principal investigator, Assiut University
Other Study IDs: Chronic hemolytic anemia
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Hemolytic Anemia, Chronic; Liver Diseases
MeSH Terms: conditions — Anemia, Hemolytic; Bronchiolitis Obliterans Syndrome; Liver Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to detect risk factors for liver affection in patients with chronic hemolytic anemias presented to the hematology unit.

DETAILED DESCRIPTION:
Hemolytic anemia is defined as decreased levels of erythrocytes in circulating blood due to their premature destruction.It is classified to acute and chronic haemolytic anemia ,chronic hemolytic anemia includes thalassemia and sickle cell anemia.

A thalassemia is a group of hereditary disorders. Mutations causing this disease reduce the production of alpha-globin and beta (β) -globin chains ,Beta thalassemia is an autosomal recessive disorder that results from genetic deficiency in the synthesis of beta-globin chains. There are more than 200 known mutations in beta globin gene that cause thalassemia thus it has wide spectrum of severity. Clinically, beta thalassemia syndromes are classified into thalassemia trait, transfusion dependent thalassemia "TDT" or non-transfusion-dependent thalassemia " NTDT

TDT" patients are liable for several medical complications that can lead to death. Liver disease is the most important and common of them. Common risk factors for this are extramedullary hematopoiesis, hepatic iron overload, infection with hepatitis virus and chelation therapy toxicity.Thalassemia traditionally has a high prevalence in the Mediterranean area, countries in the Middle East, the Arabic peninsula and Southeast Asia.

Patient with Sickle cell disease (SCD) have experienced a great amelioration in quality of life, appreciations goes to the introduction of modern transfusions of filtered red cells . However, blood transfusions cause iron accumulation over the years, and in the absence of physiologic ability to excrete excess iron , there is a progressive damage of major organs; such as the heart, the liver, and endocrine system .

Iron accumulation can be measured by determining serum ferritin levels because it best reflects the body's iron status.Liver is a storage place for iron and the only site of transferrin and ferritin synthesis, and hence the first organ to be affected.chelation therapy is necessary to prevent iron accumulation and/or to remove excess iron.

Liver involvement in patients with chronic haemolytic anemia includes a wide range of alterations, from mild liver function test abnormalities to cirrhosis and acute liver failure.the pathogenesis of cirrhosis is related to chronic hepatitis B or C infection and iron overload as a result of hemolysis and multiple transfusions that these patients require in their lifetime.

Patients with B thalassemia are at increased risk of hepatocellular carcinoma (HCC).the risk of HCC development in beta-thalassemia is linked to several factors: the high risk of infections transmitted by blood transfusions, responsible of chronic liver diseases as hepatitis C virus (HCV) and, hepatitis B virus (HBV); the debatable risk that blood transfusions inhibit immune-surveillance against cancer .

ELIGIBILITY:
Inclusion Criteria:

* All patients presented to Clinical Hematology unit, Internal Medicine Department at Assuit university University with

  * thalassemia .
  * sickle cell anemia.

Exclusion Criteria:

* patients with history of :

  * alcohol consumption
  * malignancy
  * autoimmune hepatitis

Ages: 1 Month to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: It is cross sectional descriptive study in which all patients with B thalassemia and sickle cell anemia will be included.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
To detect risk factors for liver affection in patients with chronic hemolytic anemias presented to the hematology unit. | 12/2024 - 12/2026
  Liver involvement in patients with chronic haemolytic anemia includes a wide range of alterations, from mild liver function test abnormalities to cirrhosis and acute liver failure.the pathogenesis of cirrhosis is related to chronic hepatitis B or C infection and iron overload as a result of hemolysis and multiple transfusions that these patients require in their lifetime Patients with B thalassmia are at increased risk of hepatocellular carcinoma (HCC).the risk of HCC development in beta-thalassemia is linked to several factors: the high risk of infections transmitted by blood transfusions, responsible of chronic liver diseases as HCV and, HBV; the debatable risk that blood transfusions inhibit immune-surveillance against cancer

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abbas Al masry, Pro, Study Director — Assiut University